CLINICAL TRIAL: NCT06009874
Title: Clinical Investigation of Cardioprotective Effect of Early Administration of Sodium-glucose Cotransport-2 Inhibitors in Patients With Acute Myocardial Infarction
Brief Title: Clinical Investigation of the Cardioprotective Effect of Early Administration of SGLT2 in Patients Presented With AMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammad Hussien Tantawy Soliman (Other)
Responsible Party: Sponsor-Investigator, Mohammad Hussien Tantawy Soliman, Principal Investigator, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 35541/6/22
Record Dates: First submitted 2023-08-11; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin group (Active Comparator): patients with MI will be treated with DAPA 10 mg once daily for three months.
  Interventions: Drug: Dapagliflozin 10mg Tab
- Placebo group (Placebo Comparator): patients with MI will be treated with a matching placebo once daily for three months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — patients will be treated with DAPA 10 mg once daily for three months
  Other Names: DAPA
  Arms: Dapagliflozin group
Drug: Placebo — patients will be treated with a placebo tab once daily for three months
  Arms: Placebo group

SUMMARY:
This study aims to investigate the effect of early administration of DAPA during ischemia and before pPCI on infarct size, reperfusion injury-related myocardial damage, cardioprotection from HF, and renoprotection from AKI in patients with AMI.

DETAILED DESCRIPTION:
DAPA was approved for HF patients, but there is no sufficient data about its efficacy on patients with AMI and if it can protect from the development of HF after AMI.

the investigators aim to investigate the effect of DAPA on patients who presented with AMI when administered as early as possible before pPCI and to be continued for three months after there.

the effect of DAPA on infarct size, cardiac biomarkers will be assessed during the follow-up period

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ST-elevation myocardial infarction (STEMI).
2. STEMI was defined according to the Fourth Universal Definition of AMI.
3. 18 - 80 years of age.
4. Diabetics or non-diabetics.
5. eGFR > 45 ml/min/1.73m2.
6. Blood pressure before first drug dosing >110/70 mmHg.

Exclusion Criteria:

1. Cardiogenic shock.
2. Hypoglycemia.
3. History of diabetic ketoacidosis.
4. Genital and urinary infections.
5. History of AMI.
6. Stent thrombosis.
7. Previous coronary artery bypass surgery.
8. Severe hepatic insufficiency.
9. Advanced cancer patients.
10. Blood pH < 7.32.
11. Known allergy to SGLT-2 inhibitors.
12. Hemodynamic instability.
13. Females of childbearing potential without adequate contraceptive methods.
14. Patients currently on or have received any SGLT-2 inhibitors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
difference in infarct size | 3 months
  infarct size measurement (percentage) for both groups
difference in NT-proBNP level | 3 months
  NT-proBNP level (pg/ml) for both groups

SECONDARY OUTCOMES:
Difference in eGFR | 3 months
  Decline in eGFR (ml/min) for both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Soliman, Shibīn al Kawm, Menofia, Egypt

IPD SHARING:
Plan to Share IPD: No